CLINICAL TRIAL: NCT07115095
Title: Evaluation of Serum Tumor Markers in Assessing the Efficacy of TP Chemotherapy Combined With Trastuzumab and Pertuzumab Dual Target Therapy in HER2-Positive Breast Cancer
Brief Title: Tumor Markers for Efficacy of Dual-Target Therapy in HER2+ Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanlin Li (Other)
Responsible Party: Sponsor-Investigator, Nanlin Li, Principal investigator, Shaanxi Provincial Cancer Hospital
Organization: Shaanxi Provincial Cancer Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20202039-C-1
Record Dates: First submitted 2025-07-27; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — Trastuzumab; pertuzumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Study Group (Dual-Target Therapy) (Experimental): Patients received TP chemotherapy combined with trastuzumab and pertuzumab. Treatment was administered for 6 cycles, with each cycle lasting 21 days.
  Interventions: Drug: TP Chemotherapy + Trastuzumab + Pertuzumab
- Active Comparator: Control Group (Single-Target Therapy) (Active Comparator): Patients received TP chemotherapy combined with trastuzumab only. Treatment was administered for 6 cycles, with each cycle lasting 21 days.
  Interventions: Drug: TP Chemotherapy + Trastuzumab

INTERVENTIONS:
Drug: TP Chemotherapy + Trastuzumab + Pertuzumab — Chemotherapy regimen: Paclitaxel (150 mg/m²) intravenously on Day 1 and Carboplatin (400 mg/m²) intravenously on Day 2. Targeted therapy: Trastuzumab (8 mg/kg) intravenously and Pertuzumab (initial dose 840 mg, subsequent doses 420 mg) intravenously. This regimen was repeated every 21 days for 6 cycles.
  Arms: Experimental: Study Group (Dual-Target Therapy)
Drug: TP Chemotherapy + Trastuzumab — Chemotherapy regimen: Paclitaxel (150 mg/m²) intravenously on Day 1 and Carboplatin (400 mg/m²) intravenously on Day 2. Targeted therapy: Trastuzumab (8 mg/kg) intravenously. This regimen was repeated every 21 days for 6 cycles.
  Arms: Active Comparator: Control Group (Single-Target Therapy)

SUMMARY:
This is a prospective, randomized study to compare the efficacy of TP (Taxane plus Carboplatin) chemotherapy combined with dual-HER2 blockade (trastuzumab and pertuzumab) versus TP chemotherapy plus single-HER2 blockade (trastuzumab) in patients with HER2-positive breast cancer. The study aims to evaluate treatment response and the clinical value of serum tumor markers (CEA, CA125, and CA153) in assessing therapeutic efficacy.

DETAILED DESCRIPTION:
Human epidermal growth factor receptor 2 (HER2)-positive breast cancer accounts for 15-20% of all breast cancers and is associated with a more aggressive disease course. Dual blockade of the HER2 pathway with trastuzumab and pertuzumab, in combination with chemotherapy, has become a standard of care. This study was designed to investigate the added benefit of pertuzumab to a regimen of TP chemotherapy and trastuzumab. Ninety-eight patients with HER2-positive breast cancer were randomized to receive either TP chemotherapy with trastuzumab and pertuzumab (Study Group) or TP chemotherapy with trastuzumab alone (Control Group). The primary objectives were to compare the overall response rate (ORR) and disease control rate (DCR) between the two arms. Secondary objectives included the evaluation of changes in serum tumor marker levels (CEA, CA125, CA153) before and after treatment, the predictive value of these markers for treatment efficacy, and the safety profile of the regimens.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed HER2-positive breast cancer.
* Presence of measurable lesions.
* No evidence of distant metastases.
* No prior surgery or chemotherapy.
* Voluntarily signed the informed consent form.

Exclusion Criteria:

* Incomplete neoadjuvant therapy.
* Incomplete clinical medical records.
* Presence of distant organ metastasis.
* Known allergy to study drugs.
* Expected survival of less than 3 months.
* Significant liver or kidney dysfunction.
* Presence of hematological or immune system diseases.
* Unclear pathological results.
* Concurrent other malignant tumors.
* Pregnant or lactating patients.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | After completion of Cycle 6 (each cycle is 21 days)
  The proportion of patients with a complete response (CR) or partial response (PR) according to iRECIST criteria.
Disease Control Rate (DCR) | After completion of Cycle 6 (each cycle is 21 days)
  The proportion of patients with a complete response (CR), partial response (PR), or stable disease (SD) according to iRECIST criteria.

SECONDARY OUTCOMES:
Change in Serum Carcinoembryonic Antigen (CEA) level | Baseline and after completion of Cycle 6 (each cycle is 21 days)
  Measured from serum samples. Unit: ng/mL.
Change in Serum Carbohydrate Antigen 125 (CA125) level | Baseline and after completion of Cycle 6 (each cycle is 21 days)
  Measured from serum samples. Unit: U/mL.
Change in Serum Carbohydrate Antigen 153 (CA153) level | Baseline and after completion of Cycle 6 (each cycle is 21 days)
  Measured from serum samples. Unit: U/mL.
Incidence of Treatment-Related Adverse Events | Monitored throughout the treatment period, from Baseline up to the completion of Cycle 6 (each cycle is 21 days)
  Number of participants experiencing adverse events, graded according to the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Events include liver function abnormalities, hemoglobin reduction, platelet reduction, cardiotoxicity, gastrointestinal symptoms, and joint/muscle pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China